CLINICAL TRIAL: NCT06476002
Title: Analysis of the Understanding of the French Translation of the Vulvar Pain Assessment Questionnaire (VPAQscreen) and Its Supplemental Scales (VPAQdesc, VPAQcope and VPAQpartner).
Brief Title: Analysis of the Understanding of the French Version of the Vulvar Pain Assessment Questionnaire
Acronym: VPAQ-Trad
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2023_0090
Record Dates: First submitted 2024-06-11; First posted 2024-06-26 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Vulvodynia
MeSH Terms: conditions — Vulvodynia | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- women with provoked or mixed vestibulodynia (Other): Completion of translated VPAQscreen, VPAQdesc, VPAQcope and VPAQpartner questionnaires by patients, followed by assessment of comprehension of the various items.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Completion of translated VPAQscreen, VPAQdesc, VPAQcope and VPAQpartner questionnaires by patients, followed by assessment of comprehension of the various items.

SUMMARY:
Prior to the current study, a translation into french of the screening version of the VPAQ (VPAQscreen) and its supplemental scales (VPAQdesc, VPAQcope, VPAQpartner) was performed according to the recommended process. The present study aims to evaluate the understanding of this translation on a panel of 30 women suffering from provoked or mixed vestibulodynia.

DETAILED DESCRIPTION:
The Vulvar Pain Assessment Questionnaire (VPAQ) is a self-assessment questionnaire for chronic vulvar pain. The English-language version has been validated on patients suffering from chronic pain of various causes, mainly vulvodynia. It explores the biopsychosocial dimensions of chronic vulvar pain: description, intensity, temporality, associated symptoms, emotional and cognitive functioning, coping strategies and interpersonal relations with the partner. The VPAQ inventory is divided into a main questionnaire (VPAQfull or a shorter version, VPAQscreen) and 3 supplementary questionnaires exploring Pain Descriptors (VPAQdesc), coping strategies (VPAQcope) and partner factors (VPAQ partner). The VPAQ inventory can be used both for research purposes and clinical practice. Indeed, it helps the patients to better express their symptoms and the providers to cover with one tool all the dimensions of chronic vulvar pain. A french translation would make the VPAQ inventory available for french speaking health care professionals and patients.

The aim of our study is to validate a french translation of the VPAQscreen and its three supplementary questionnaires. Prior to this study, a french translation of these questionnaires was performed according to the recommended process.

Whereas the English VPAQ inventory has been validated on patients with chronic vulvar pain, whatever the cause, the investigators have chosen to carry out this validation on a homogeneous population of women suffering from provoked or mixed vestibulodynia (i.e, pain located on the vulvar vestibule, triggered by local contacts and associated or not with spontaneous pain). Indeed, provoked vestibulodynia is the most frequent and the best-defined clinical subset of vulvodynia (i.e, chronic vulvar pain with no identifiable cause). The investigators excluded patients suffering from vulvodynia involving other sites than the vestibule as well as chronic vulvar pain related to specific causes (neurological, myofascial, etc..) The understanding of this french translation of the VPAQ will be tested on a panel of 30 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* with a diagnosis of provoked or mixed vestibulodynia confirmed by an expert gynecologist or vulvar dermatologist
* Have signed a consent form
* French mother tongue and able to read
* Affiliated to a social security scheme

Exclusion Criteria:

* Patient with vulvar pain associated with other pathologies
* Deprived of liberty or under guardianship.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2024-05-06 (Actual); Primary Completion 2025-02-06 (Actual); Study Completion 2025-02-06 (Actual)

PRIMARY OUTCOMES:
understanding question | Day 1
  for each item of VPAQscreen (Vulvar Pain Assessment Questionnaire Screen) and the specific supplementary questionnaires (VPAQdesc, VPAQcope, VPAQpartner), answer to "Did you understand that question?"
understanding answer | Day 1
  for each item of VPAQscreen (Vulvar Pain Assessment Questionnaire Screen) and the specific supplementary questionnaires (VPAQdesc, VPAQcope, VPAQpartner), answer to "Did you understand the different possible answers?"
understanding | Day 1
  for each item of VPAQscreen (Vulvar Pain Assessment Questionnaire Screen) and the specific supplementary questionnaires (VPAQdesc, VPAQcope, VPAQpartner), answer to "Can you explain what went wrong?"

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Foch, Suresnes, France

IPD SHARING:
Plan to Share IPD: No